CLINICAL TRIAL: NCT06665854
Title: Effect of Rhythm Therapy on Fetal Learning, Prenatal Attachment and Prenatal Distress in Pregnant Women
Brief Title: Effect of Rhythm Therapy Practices on Fetal Learning, Prenatal Attachment and Prenatal Distress
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAU-SBF-BNYB-01
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Prenatal Attachment; Prenatal Stress; Fetal Outcomes
Keywords: Prenatal Attachment; Prenatal Stress; Fetal Learning; Primiparous Pregnancy; Rhythm Therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: After reaching the sample number of pregnant women for this study, pregnant women will be assigned to groups as group 1, group 2, and control group by block randomization method. This method will be used to eliminate selection bias and ensure balance between groups in terms of individuals. Random numbers table will be used in the selection of pregnant women.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rhythmic Song Group (Experimental): The rhythmic song group will ring a bell when starting to stimulate the baby, and will code the baby's movements as present/absent via the mobile application; then it will sing a rhythmic song and code the baby's movements as present/absent via the mobile application again.
  Interventions: Behavioral: Rhythmic Song Group
- Rhythmic Instrument Group (Experimental): The Rhythmic Instrument Group will ring a bell when starting the application to stimulate the baby, and will code the baby's movements as present/absent via the mobile application; then they will play a rhythmic instrument and code the baby's movements as present/absent via the mobile application again.
  Interventions: Behavioral: Rhythmic Instrument Group
- Control Group (Placebo Comparator): The control group will ring a bell to warn the baby, they will code the baby's movements as present/absent via the mobile application again, and they will only rest.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Rhythmic Song Group — The rhythmic song group will first click on the start button on the mobile application. When starting the application to stimulate the baby, a bell will ring, and the baby movements will be coded as present/absent via the mobile application; then they will sing a rhythmic song and recode the baby movements as present/absent via the mobile application. Applications will begin in the 28th week of pregnancy and continue until the 37th week of pregnancy. Pregnant women will receive rhythm therapy applications for 20 minutes twice a week.
  Arms: Rhythmic Song Group
Behavioral: Rhythmic Instrument Group — The Rhythmic Instrument Group will first click on the start button on the mobile application. Then, they will ring a bell to start the application to warn the baby, and they will code the baby's movements as present/absent via the mobile application; then they will play a rhythmic instrument and code the baby's movements as present/absent via the mobile application again. Applications will begin in the 28th week of pregnancy and continue until the 37th week of pregnancy. Pregnant women will receive rhythm therapy applications for 20 minutes twice a week.
  Arms: Rhythmic Instrument Group
Behavioral: Control Group — Control Group will first code "Start" via the mobile application. Then, a bell will ring to warn the baby, they will code the baby's movements as present/absent via the mobile application again and will only rest. When the application is over, all pregnant women will code "Finish" via the mobile application. Applications will begin in the 28th week of pregnancy and continue until the 37th week of pregnancy. Pregnant women will receive rhythm therapy applications for 20 minutes twice a week.
  Arms: Control Group

SUMMARY:
The concept of prenatal attachment defines the relationship between the pregnant woman and the foetus. The attachment established between the mother and the baby is an important factor in the quality of care and survival of the baby in the postnatal period, and the quality of the interaction established with the mother is also a determinant of the cognitive and social development of the baby. One of the factors affecting prenatal attachment is the stress factor. Stress also affects foetal life and has negative consequences in many life stages including neonatal period, childhood and adulthood. Another factor affecting prenatal attachment is foetal learning, which is defined as the process of intrauterine memory development. Within the scope of this study, rhythm therapy and music applications based on rhythm applications and mother's voice will be used. The effects of rhythm therapy during pregnancy on fetal learning, prenatal stress, prenatal attachment and neonatal outcomes will be examined in this study. In addition, within the scope of the study, a mobile application will be developed and installed on the phones of pregnant women and the processes related to fetal learning will be monitored online through this application. The study was planned as a randomised controlled study. All pregnant women who agree to participate in the study will first be administered the descriptive characteristics form, prenatal attachment and prenatal stress scales. Then, online trainings about the topics included in the study will be given and a mobile application will be installed on their phones. Pregnant women will be divided into 3 groups; pregnant women in the 1st group will be taught rhythmic song writing, pregnant women in the 2nd group will be taught to play rhythmic instruments and the 3rd group will be determined as the control group. The women will apply rhythmic music applications to the foetus for 20 minutes every 2 days for 2 days every week until the birth and will make coding through the mobile application installed on their phones. The response of the fetus to the music applications will be evaluated through fetal movements. At 37 weeks of gestation, prenatal attachment and prenatal stress scales will be applied and the effect of music applications will be evaluated. In this way, the effects of music practices applied in the fetal period on fetal memory, prenatal attachment and prenatal stress will be evaluated at the same time. A study of this type has not yet been found in the domestic and foreign literature. In addition, the use of mobile application within the scope of the study will contribute to the literature on mobile health applications.

DETAILED DESCRIPTION:
The proposed project has been transferred as 2 main Work Packages (WP). WP 1. Shooting of training videos. WP 2. Investigation of the effect of rhythm therapy application in pregnant women on prenatal attachment, prenatal stress and fetal learning.

Mobile application: A mobile application specific to the project has been developed for use by the project manager. There are 5 interfaces in this mobile application. The first interface contains the login information of the pregnant women (name-surname-gestational week-email address). Pregnant women will register to the application through this interface and their gestational age will be monitored. In this way, the manager will track the gestational week in which the applications made by the participants were made during the data collection phase of the project. The second interface contains the Socio-Demographic Characteristics Form, Prenatal Attachment Inventory and Prenatal Stress Scale to be filled out by pregnant women within the scope of the project. Pregnant women will fill out these forms at the latest at the 27th week of pregnancy before starting data collection. The third interface contains the training videos to be used in the research. Participants will complete the training videos at the latest by the 27th week of pregnancy before starting the data collection phase. The fourth interface contains the pregnancy period coding section. With the coding section in this interface, participants will code the fetal movements during rhythm therapy applications. The fifth intermediary includes the Prenatal Attachment Inventory and Prenatal Stress Scale to be filled out at the 37th week of pregnancy. Each interface is designed to be conditional on each other. Participants will follow the steps in each interface in order.

There are two main purposes for using this mobile application in this project. The first purpose is to use it during the pregnancy data collection phase of the project. Within the scope of this project, participants will be able to easily enter data through the mobile application while performing rhythm therapy applications. Thanks to the main screen loaded onto the manager's computer, it will be possible to track when rhythm therapy and music applications are performed and whether there are any baby movements after the application, thanks to the coding. In addition, thanks to the mobile application, pregnant women and postpartum mothers will be able to easily participate in the study in their own environment without coming to the hospital. This is a cost-effective method and provides opportunities for both the manager and the participants in terms of time management. The researcher will be able to follow the study data through the interface on his/her computer.

Work Package 1. Shooting of training videos: Two groups of videos will be shot within the scope of the project. The first group of videos will be on rhythm therapy. Within the scope of the project, pregnant and postpartum women are expected to write rhythmic songs/lullabies and play rhythmic instruments. The project manager has received Theoretical 3 (Distance Education) / Practical 1 (Distance Education) - Total: 4 weeks training from the Republic of Turkey Rhythm Therapy Music and Rhythm Therapy Education-Research and Application Center and has earned the right to receive a Rhythm Therapist Certificate. In addition, he/she has completed the 40-hour Music Therapy and Awareness Raising Training conducted by the Sakarya University of Applied Sciences Lifelong Education Application and Research Center and has earned the right to receive a certificate. Training videos on rhythm therapy will be shot by the project manager for the participants and will be shared with the participants who volunteer to participate in the project via the mobile application before data collection. There will be 2 videos in the first group. The subject of the first video has been determined as Music and Rhythm Therapy, and the subject of the second video has been determined as Writing rhythmic songs/lullabies and playing rhythmic instruments (metal xylophone). All videos will be shot by the facilitator at Sakarya Education and Research Hospital. The second group of videos will be videos specific to the application. Sample videos will be shot to provide information and reference to the participants during the pregnancy data collection phase of the project. 3 groups will be formed during the data collection phase of this project. These videos will include applications specific to the groups. Group 1 is the Rhythmic Song Group, Group 2 is the Rhythmic Instrument Group and Group 3 is the Control Group. During the data collection phase of the study, each group will apply the intervention specific to their group. Pregnant women will not have a need to urinate at the time of the application, they will be full and they will prefer a quiet and calm room for the application. No physical stimulation will be given to the abdomen during the application and a resting position will be taken. All pregnant women will code "Start" via the mobile application when starting. Pregnant women in the first group (rhythmic song group) will ring a bell to stimulate the baby and code the baby movements as present/absent via the mobile application; then they will sing a rhythmic song and code the baby movements as present/absent via the mobile application again. The second group of pregnant women (Rhythmic Instrument Group) will ring a bell to stimulate the baby, code the baby movements as present/absent via the mobile application; then play a rhythmic instrument and code the baby movements as present/absent via the mobile application again. The third group (control group) will ring a bell to stimulate the baby, code the baby movements as present/absent via the mobile application again and will only rest. When the application is over, all pregnant women will code "Finish" via the mobile application. A reference video will be shot to ensure that all these application patterns are more permanent in the minds of the pregnant women. The video pattern will be prepared by the facilitator and the shots will be made so that the intervention steps are clearly visible. These videos will be specific to each group and will be integrated into the mobile application and easily accessible.

Work Package 2. Investigation of the effects of rhythm therapy applications on prenatal attachment, prenatal stress and fetal learning in pregnant women:

Type of research: The research was planned as a randomized control group intervention study with a pretest-posttest design from fully experimental research designs. This study will be reported in accordance with the CONSORT guideline.

Research universe and sample: The universe of the proposed project consists of pregnant women who meet the inclusion and exclusion criteria and apply to the Sakarya Education and Research Hospital Birth Preparation Class and healthy pregnancy polyclinic. The sample of the research was determined by power analysis. As a result of the power analysis applied with the power analysis 3.1.9.7 program, the sample size was determined as 22 people in the groups and 66 people in total according to the value of type 1 error: 0.05, type 2 error: 0.20 and effect size = 0.40 for the determination of differences in measurements between the groups. Considering the situation calculated due to possible losses in the study, the sample size was increased by 20% and it was planned to include 78 people, 26 in each group.

Inclusion, Exclusion and Exclusion criteria for the study:

Inclusion Criteria: Agreeing to participate in the study, Knowing Turkish, Being a primiparous pregnancy, Not being a high-risk pregnancy, Being a singleton pregnancy, Being between 20 and 27 weeks of gestation.

Exclusion Criteria: Being pregnant with assisted reproductive techniques, Not using a smart phone.

Exclusion Criteria: Not performing rhythm therapy applications twice a week, Not coding during rhythm therapy applications, Leaving the study, Giving birth earlier than the expected date, The baby staying in the neonatal intensive care unit during the first week after birth.

Randomization:

After reaching the number of pregnant women for the project, the pregnant women will be assigned to the groups as group 1, group 2 and the control group with the block randomization method. This method will be used to eliminate selection bias and ensure balance between groups in terms of individuals. A random number table will be used in the selection of pregnant women.

Data collection tools:

A mobile application will be installed on the phones of participants who agree to participate in the study. The Socio-Demographic Characteristics Form, Prenatal Attachment Inventory and Prenatal Distress Scale integrated into the mobile application will be filled out by all pregnant women as a pre-test and post-test.

Implementation of the research:

Choosing the Rhythmic Musical Instrument: It is known that the music that the fetus is exposed to during the fetal period has fluent and soft melodies and a heart rate of 60-80 beats/min, similar to the human heart rate, affects fetal hearing. It is thought that the beat rate compatible with the maternal heart rate strengthens the learning of babies, as stated in the studies. For this purpose, the Metal Xylophone was selected as the rhythmic musical instrument in the proposed project.

Within the scope of the project, groups will be formed with randomization and after the pre-test application is completed, the phase of providing rhythm training will be started. At this stage, the theoretical trainings on Music and Rhythm Therapy and Writing Rhythmic Songs/Lullabies and Playing Rhythmic Instruments, which were previously shot by the researcher and uploaded to the mobile application, will be completed by the participants. Online trainings on writing rhythmic songs/lullabies and playing rhythmic instruments will be carried out by making appointments with the participants who have completed their theoretical trainings. After these trainings are completed, the practices that Group 1 (Rhythmic Song Group) and Group 2 (Rhythmic Instrument Group) will apply during pregnancy and postpartum will be determined for the data collection phase. Pregnant women will apply the intervention of the group they are assigned to for 20 minutes twice a week starting from the 3rd trimester (28th week). Before the rhythm therapy applications, all pregnant women in the group will be told that they should not have any urinary urgency, that they should be full, that the environment should be quiet, calm, at an appropriate temperature and that it should support mother-fetus interaction, and that they should not touch their abdomens during the intervention.

During the data collection phase of the study, a post-test will be applied to all pregnant women who have reached the 37th week of pregnancy and are included in the study. The Prenatal Attachment Inventory and Prenatal Distress Scale integrated into the mobile application will be applied again in the post-test application. As a result of the statistical interpretation of the pre-test and post-test applications, the effect of rhythm therapy applications on prenatal attachment and prenatal stress will be investigated. In order to carry out the proposed project, an ethics committee permit (dated 14.11.2023 and numbered E16214662-05.01.04-305616) was obtained from Sakarya University.

Data analysis:

The data in the study will be completed by transferring them to the International Business Machines Statistical Package for the Social Sciences Statistics 26 program. When evaluating the study data, frequency distribution (number, percentage) will be given for categorical variables and descriptive statistics (mean, standard deviation, median, minimum, maximum) will be given for numerical variables. One-way analysis of variance (One Way ANOVA) will be used for variables that are normally distributed, and Kruskal Wallis test will be used for variables that are not normally distributed. In addition, dependent sample t-test will be used for variables that are normally distributed, Wilcoxon test will be used for variables that are not normally distributed, and Cronbach alpha value will be used for scale reliability to examine the change in measurements over time. P<0.05 will be accepted as significance.

ELIGIBILITY:
Inclusion Criteria:

Accepting to participate in the study, Knowing Turkish, Being a primiparous pregnancy, Not being a high-risk pregnancy, Being a singleton pregnancy, Being between 20 and 27 weeks of gestation.

Exclusion Criteria:

Not performing rhythm therapy applications twice a week, Not coding during rhythm therapy applications, Leaving the study, Giving birth before the expected date.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Socio-Demographic Characteristics Form | 27th week of pregnancy
  It was created by the researchers and contains 18 questions covering the socio-demographic characteristics of the participants.
Prenatal Attachment Inventory | 27th week of pregnancy and 38th week of pregnancy
  It is a 21-item inventory developed by Mary Muller (1993) to explain the thoughts, feelings, and situations experienced by women during pregnancy and to determine the level of attachment to the baby in the prenatal period. It was adapted to Turkish in Turkey in 2010 and the Cronbach alpha reliability coefficient was found to be 0.84. It has been suggested that the Prenatal Attachment Inventory is a valid and reliable tool for pregnant women in our country and that it can be used by researchers in studies to determine the level of attachment of pregnant women with different characteristics to their babies in the prenatal period.
Prenatal Distress Scale | 27th week of pregnancy and 38th week of pregnancy
  It was first developed in 1999 to assess specific concerns and anxieties specific to pregnancy, such as medical problems, physical symptoms, parenting, relationships, physical changes, birth, and the baby's health. It was adapted to Turkish in 2011, and the Cronbach alpha internal consistency coefficient was found to be 0.85. It was determined that the Turkish form of the Prenatal Distress Scale is an understandable, valid, and reliable tool for use on Turkish pregnant women in the assessment of stress that may occur during pregnancy in our country.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Nur Yıldırım Bayraktar, PhD Candidate, Study Director — Sakarya University; Kevser İlçioğlu, Associate professor, Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want my data to be shared.